CLINICAL TRIAL: NCT05435885
Title: Comparison of Postoperative Telerehabilitation and Unsupervised Home-Based Training in Older Adults With Lung Cancer: A Randomized Controlled Trial
Brief Title: Postoperative Telerehabilitation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2205-033-114
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Telerehabilitation; Carcinoma, Non-Small-Cell Lung; Cardiopulmonary Exercise Test
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation group (Experimental): The Tele-rehabilitation group performs 12 training sessions during four weeks. (3 sessions/week)
  Interventions: Other: Pulmonary Tele-Rehabilitation
- Control group (Other): The control group receives usual care with only one educational session.
  Interventions: Other: Control (Education)

INTERVENTIONS:
Other: Pulmonary Tele-Rehabilitation — 12 supervised training sessions via a specific mobile messenger during four weeks. (3 sessions/week)
  Arms: Tele-rehabilitation group
Other: Control (Education) — Usual care with only one educational session.
  Arms: Control group

SUMMARY:
The purpose of this study is to confirm the effectiveness of a mobile messenger-based home tele-rehabilitation protocol in patients who have undergone lung resection surgery.

By analyzing the difference from the existing postoperative pulmonary rehabilitation, the investigators would like to propose a new pulmonary tele-rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

1. A person who is suspected of lung cancer and is scheduled to undergo a thoracoscopic lung resection surgery.
2. men and women the age ≥65 years.
3. A person who understands the course of the clinical trial and signs the informed consent form.

Exclusion Criteria:

1. Patients whose activity is restricted due to other diseases (e.g. osteoarthritis, spinal disease, cerebral infarction, etc.)
2. Patients who cannot test bioimpedance analysis due to the insertion of artificial pacemakers and defibrillators
3. A person who has difficulty judging himself/herself due to dementia, etc
4. Those enrolled in other clinical trials
5. A person deemed inappropriate to participate in this clinical trial under the judgement of the investigator.
6. A person who cannot use mobile messenger

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hun Kim, M.D.,Ph.D., Study Director — Pusan National University Hospital
Locations (1):
- PusanNUH, Pusan, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 96 participants were assessed for eligibility. Of these, 64 were randomized.
Period: Overall Study
Arm/Group | Tele-rehabilitation Group | Control Group
Started | 29 | 35
Completed | 26 | 33
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-rehabilitation Group | Control Group | Total
Number analyzed (Participants) | 29 | 35 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 29 | 35 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (5) | 72.2 (5) | 71.9 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 15 | 21 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 29 | 35 | 64
BMI [Mean (Standard Deviation); unit: kg/m2] | 24 (3) | 24 (4) | 24 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in VO2 Peak (Peak Oxygen Uptake, mL/kg/Min) on the CardioPulmonary Exercise Test(CPET) After 4 Weeks Intervention
Description: Cardiopulmonary exercise test (CPET) also referred to as a VO2 (oxygen consumption) test, is a specialized type of stress test or exercise test that measures participants exercise ability.
Time Frame: Before surgery (Pre), Baseline (4 weeks after surgery), After intervention(8 weeks after surgery), Follow up(12 weeks after surgery)
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
mL/kg/min
  Before surgery (Pre) | 23.67 (4.64) | 23.09 (4.73)
  Baseline (4 weeks after surgery) | 19.28 (4.16) | 20.41 (3.62)
  After intervention(8 weeks after surgery) | 21.85 (4.22) | 19.85 (4.02)
  Follow up(12 weeks after surgery) | 21.73 (4.18) | 19.82 (3.89)

2. Secondary Outcome: Ventilatory Efficiency (VE/VCO₂ Slope)
Description: VE/VCO₂ slope measured during CPET. Lower values indicate better ventilatory efficiency.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
ratio
  Within-Group Differences in VE/VCO₂ Slope Immediately After Rehabilitation | 4.0 [1.1 to 6.9] | 0.6 [-3.0 to 4.2]
  Within-Group Differences in VE/VCO₂ Slope at 4-Week Follow-Up | -0.1 [-2.5 to 2.4] | 1.4 [-1.4 to 4.2]

3. Secondary Outcome: Maximal Inspiratory Pressure (MIP)
Description: Maximal inspiratory pressure measured using a handheld respiratory device. Higher values indicate stronger inspiratory muscles. Unit of Measure: cmH₂O
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: cm/H2O
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
cm/H2O
  Within-Group Differences in Maximal Inspiratory Pressure Immediately After Rehabilitation | 5.2 [-2.2 to 12.6] | 8.3 [3.8 to 12.9]
  Within-Group Differences in Maximal Inspiratory Pressure at 4-Week Follow-Up | 7.9 [0.4 to 15.4] | 5.4 [-1.4 to 12.1]

4. Secondary Outcome: Skeletal Muscle Index (SMI)
Description: Skeletal muscle index calculated by dividing appendicular skeletal muscle mass by height squared. Higher values indicate greater muscle mass.
  Unit of Measure: kg/m²
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: kg/m²
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
kg/m²
  Within-Group Differences in Skeletal Muscle Index Immediately After Rehabilitation | 0.1 [-0.2 to 0.3] | -0.1 [-0.6 to 0.3]
  Within-Group Differences in Skeletal Muscle Index at 4-Week Follow-Up | 0.1 [-0.01 to 0.2] | 0.11 [0.01 to 0.2]

5. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) was devised 30 years ago by Zigmond and Snaith to measure anxiety and depression in a general medical population of patients.
  The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression.
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
score on a scale
  Within-Group Differences in HADS Anxiety Score Immediately After Rehabilitation | -0.4 [-1.8 to 1.1] | 0.6 [-0.5 to 1.8]
  Within-Group Differences in HADS Anxiety Score at 4-Week Follow-Up | -0.9 [-2.2 to 0.4] | -0.1 [-1.0 to 0.8]
  Within-Group Differences in HADS Depression Score Immediately After Rehabilitation | -1.1 [-2.4 to 0.2] | -0.6 [-1.9 to 0.7]
  Within-Group Differences in HADS Depression Score at 4-Week Follow-Up | -1.0 [-2.5 to 0.5] | -1.2 [-2.5 to 0.1]

6. Secondary Outcome: EQ-5D (EuroQol-5 Dimension)
Description: The EQ-5D-5L is a standardized instrument developed by the EuroQol Group to measure health-related quality of life. It consists of two parts: a descriptive system and a visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels:
  (1) no problems, (2) slight problems, (3) moderate problems, (4) severe problems, and (5) extreme problems.
  Responses are converted into a summary index score, which ranges from -0.281 to 1.000, based on country-specific value sets. Higher index scores indicate better health status, with 1.000 representing full health and values below 0 indicating health states considered worse than death.
  The EQ VAS records the participant's self-rated health on a vertical visual analogue scale ranging from 0 to 100, where 100 represents the best health imaginable and 0 represents the worst health imaginable.
  Higher VAS scores reflect
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
score on a scale
  Within-Group Differences in EQ-5D-5L Index Score Immediately After Rehabilitation | 0.05 [0.01 to 0.10] | -0.03 [-0.07 to 0.01]
  Within-Group Differences in EQ-5D-5L Index Score at 4-Week Follow-Up | 0.05 [-0.01 to 0.10] | 0.0 [-0.05 to 0.04]
  Within-Group Differences in EQ-5D-5L Visual Analog Scale Score Immediately After Rehabilitation | 6.4 [0.3 to 12.4] | 5.4 [-0.3 to 11.0]
  Within-Group Differences in EQ-5D-5L Visual Analog Scale Score at 4-Week Follow-Up | 7.9 [0.7 to 15.1] | 7.7 [2.3 to 13.1]

7. Secondary Outcome: Grip Strength
Description: Grip strength is a measure of muscular strength or the maximum force/tension generated by participant's forearm muscles using the Jamar Hydraulic Hand Dynamometer.
  The force has been measured in kilograms.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: Kg
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
Kg
  Within-Group Differences in Grip Strength Immediately After Rehabilitation | -0.3 [-1.6 to 0.9] | 0.1 [-0.9 to 1.2]
  Within-Group Differences in Grip Strength at 4-Week Follow-Up | -0.7 [-2.3 to 0.8] | -0.2 [-1.3 to 0.9]

8. Secondary Outcome: Steps
Description: As a physical activity, Counting participant's steps per a day with an activity tracker.
  Average number of steps per day for one week before surgery and after discharge.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: steps/day
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
steps/day
  Within-Group Differences in Daily Step Count Immediately After Rehabilitation | -45 [-1090.4 to 1000.4] | -469 [-1605.5 to 666.7]
  Within-Group Differences in Daily Step Count at 4-Week Follow-Up | 1050 [-540.1 to 2640.6] | 95 [-1147.7 to 1337.7]

9. Secondary Outcome: Peak Expiratory Flow (PEF)
Description: The peak expiratory flow (PEF) is a participant's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a participant's ability to breathe out air. It measures the airflow through the bronchi and thus the degree of obstruction in the airways. Peak expiratory flow is typically measured in units of liters per minute (L/min).
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
L/min
  Within-Group Differences in Peak Expiratory Flow Immediately After Rehabilitation | 14.2 [-14.8 to 43.2] | 27.4 [3.8 to 51.0]
  Within-Group Differences in Peak Expiratory Flow at 4-Week Follow-Up | 28.7 [12.4 to 45.0] | 24.1 [6.0 to 42.2]

10. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the maximum amount of air a participant can forcibly exhale from lungs after fully inhaling.
  The unit is expressed in liters.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
Liter
  Within-Group Differences in Forced Vital Capacity Immediately After Rehabilitation | 0.17 [0.08 to 0.24] | 0.18 [0.10 to 0.26]
  Within-Group Differences in Forced Vital Capacity at 4-Week Follow-Up | 0.25 [0.13 to 0.37] | 0.23 [0.13 to 0.33]

11. Secondary Outcome: The Forced Expiratory Volume in 1 Second (FEV1)
Description: The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
Liter
  Within-Group Differences in Forced Expiratory Volume in 1 Second Immediately After Rehabilitation | 0.14 [0.07 to 0.21] | 0.11 [0.06 to 0.16]
  Within-Group Differences in Forced Expiratory Volume in 1 Second at 4-Week Follow-Up | 0.19 [0.09 to 0.28] | 0.15 [0.07 to 0.23]

12. Secondary Outcome: Whole-Body Phase Angle
Description: Bioelectrical impedance analysis (BIA)-derived phase angle (PA) is an alternative method to assess mortality risk. BIA is a simple, non-invasive technique that estimates body composition by measuring the opposition (impedance) to an applied current while passing through the body. Impedance consists of two components: resistance, which is the opposition to the flow of an alternating current through intra- and extracellular ionic solutions, and reactance, which is the delay in conduction as a result of capacitance by cell membranes and tissue interfaces.
  PA is regarded as a biological marker of cellular health, as it reflects cell mass, membrane integrity, and hydration status. PA has repeatedly proven to be a predictor of morbidity and mortality in various patient groups.
Time Frame: Immediately After Rehabilitation and at 4-Week Follow-Up
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Tele-rehabilitation Group | Control Group
Number analyzed (Participants) | 29 | 35
degrees
  Within-Group Differences in Whole-Body Phase Angle Immediately After Rehabilitation | 0.04 [-0.09 to 0.16] | -0.1 [-0.26 to 0.05]
  Within-Group Differences in Whole-Body Phase Angle at 4-Week Follow-Up | -0.02 [-0.17 to 0.13] | -0.12 [-0.29 to 0.05]

ADVERSE EVENTS:
Time Frame: Through 12 Weeks After Surgery
Description: No adverse events were reported during the study period up to 12 weeks after surgery.
Arm/Group | Tele-rehabilitation Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT05435885/Prot_SAP_000.pdf